CLINICAL TRIAL: NCT01560091
Title: Differential Effect of Silodosin Versus Tamsulosin on Stone Clearance After ESWL
Brief Title: Differential Effect of Silodosin Versus Tamsulosin on Stone Clearance After Extra-corporeal Shock Wave Lithotripsy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: accrual of subjects did not occur as anticipated
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Richard Harkaway, PRINCIPAL INVESTIGATOR, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN 4378
Record Dates: First submitted 2012-03-16; First posted 2012-03-22 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Kidney Stones
Keywords: clearance rate
MeSH Terms: conditions — Kidney Calculi | interventions — silodosin; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): Patients will receive ESWL and no medication
  Interventions: Procedure: Extra-corporeal shock wave lithotripsy
- Group B (Active Comparator): Patients will receive Flomax after ESWL
  Interventions: Procedure: Extra-corporeal shock wave lithotripsy; Drug: Tamsulosin
- Group C (Active Comparator): Patients will receive silodosin after ESWL
  Interventions: Drug: silodosin; Procedure: Extra-corporeal shock wave lithotripsy

INTERVENTIONS:
Drug: silodosin — 8mg PO Qday
  Arms: Group C
Procedure: Extra-corporeal shock wave lithotripsy — ESWL
Drug: Tamsulosin — Tamsulosin 0.4mg PO Qday
  Arms: Group B

SUMMARY:
Tamsulosin is an alpha blocker usually prescribed for urinary complaints that has been shown to have some benefit in allowing kidney stones to pass through the ureter. Silodosin is a new alpha blocker that acts more rapidly than tamsulosin and has been shown to have specific receptors on the ureter. The investigators would like to see if there is some benefit to taking silodosin over tamsulosin after extra-corporeal shock wave lithotripsy (ESWL) to break kidney stones in terms of allowing the ureteral fragments to pass through the ureter. Our hypothesis is that silodosin will be at least as effective as tamsulosin in terms of allowing stones to pass, but may allow them to pass more quickly because of the rapid onset of action.

The side effect profile for both drugs is quite similar and tolerable. Patients may experience some common side effects associated with tamsulosin, including abnormal ejaculation, dizziness, rhinitis (runny nose, sneezing), and somnolence (sleepiness). Serious reactions include orthostatic hypotension, syncope (fainting), and priapism (prolonged undesired erection).

Patients may experience some common side effects with both silodosin and tamsulosin including ejaculatory dysfunction, dizziness, postural hypotension, diarrhea, and headache. Serious side effects are rare and include orthostatic hypotension, intra-operative floppy iris syndrome, syncope, and priapism.

Patients will experience the discomfort normally associated with kidney stones. All efforts will be made to alleviate these discomforts, including the use of the study medications. Patients will be able to take their routine prescribed pain medications, and will be asked to keep a record of their pain medication use.

The investigators will be randomly enrolling patients from all racial backgrounds and of both genders. They must have kidney stones ranging in size from 4mm to 1.0 cm and have no prior treatment for the study.

The primary endpoint of this study is the clearance rate of kidney stones. That is, in what period of time does the patient achieve clearance, is stone free and has all residual stones gone. The secondary endpoints of this study include analgesic use, residual stones remaining, need for re-treatment, need for intervention, steinstrasse clearance, and the need for hospitalization.

DETAILED DESCRIPTION:
A comparison between two commonly used alpha blockers to determine if there is superiority in the secondary usage of aiding in stone passage

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 70
* Non-diabetics
* White blood cell count and serum creatinine level within normal range
* Urine analysis consistent with absence of infection
* Negative urine culture
* Absence of subjective or objective fever
* Ability to tolerate oral fluids and pain medication
* Unilateral ureteral calculus < 10mm visible on CT scan within the ureter
* Ability to make informed medical decisions regarding consent
* Willingness to follow up in the urology office

Exclusion criteria:

Adults unable to consent

* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Prior treatment for this particular stone
* Medical therapy only for stone disease
* Chronic narcotic use
* Current alpha blocker therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clearance rate of kidney stones (days) | 1 year
  The primary endpoint of this study is the clearance rate of kidney stones. That is, in what period of time does the patient achieve clearance, is stone free and has all residual stones gone. This outcome measure will be measured in days.

SECONDARY OUTCOMES:
Analgesic use | 1 year
  Analgesic use, number of pills of pain medication
Residual stones remaining | 1 year
  Residual stones remaining, based on imaging
need for re-treatment | 1 year
  need for re-treatment. Either the patient will need another ESWL, or hospitilization
need for intervention | 1 year
  need for intervention. Either ESWL again or hospitilization and further procedures such as laser lithotripsy, percutaneous nephrolithotomy, open surgery
steinstrasse clearance | 1 year
  steinstrasse clearance. Whether or not stone clearance is achieved or not
need for hospitalization | 1 year
  need for hospitalization. either yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Richard Harkaway, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided